CLINICAL TRIAL: NCT06602362
Title: Uncovering the Acute Neurobiological Significance of Emerging Sexual Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 23297
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-10

CONDITIONS: Sexual Behavior; Hypoxia, Brain
Keywords: Sexual choking
MeSH Terms: conditions — Sexual Behavior; Hypoxia, Brain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The primary investigator will be blinded to the study participants' study group status, and the statistician will be blinded from group assignment. Additionally, participants will be blinded to their own group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Path 1 (choking involved sex prior to non-choking involved sex) (Experimental): Path 1 will involve 3 data collection time points including baseline data collection, post choking involved sex data collection time point, and post non-choking involved sex time point, in that order. After enrollment, subjects will be sent a brief Qualtrics survey link once a day to determine when they are eligible for data collection based on their sexual activity within the last 24 hours. Subjects placed in the group following Path 1 will first come in for a baseline data collection which will occur after a 48 hour washout period of not engaging in partnered sex. Next, subjects will be asked to come in for an experimental data collection visit within the 24 hours post engaging in choking involved sex. Last, subjects will be asked to come in for an experimental data collection visit within 24 hours of engaging in sex that did not involve any choking.
  Interventions: Other: Partnered sex involving choking; Other: Partnered sex not involving choking
- Path 2 (non-choking involved sex prior to choking involved sex) (Experimental): Path 2 will involve 3 data collection time points including baseline data collection, post non-choking involved sex time point, and post choking involved sex time point, in that order. After enrollment, subjects will be sent a brief Qualtrics survey link once a day to determine when they are eligible for data collection based on their sexual activity within the last 24 hours. Subjects placed in the group following Path 2 will first come in for a baseline data collection which will occur after a 48 hour washout period of not engaging in partnered sex. Next, subjects will be asked to come in for an experimental data collection visit within the 24 hours after engaging in sex that did not involve any choking. Last, subjects will be asked to come in for an experimental data collection visit within 24 hours of engaging in choking involved sex.
  Interventions: Other: Partnered sex involving choking; Other: Partnered sex not involving choking

INTERVENTIONS:
Other: Partnered sex involving choking — When a subject submits a survey indicating that they engaged in partnered sex involving choking, they will be asked to come in for data collection within 24 hours of survey submission.
Other: Partnered sex not involving choking — When a subject submits a survey indicating that they engaged in partnered sex that did not involve any choking, they will be asked to come in for data collection within 24 hours of survey submission.

SUMMARY:
The purpose of this study is to examine the acute effect of being choked during partnered sex on neurological measures. The study is designed to identify the effects being choked during partnered sex on the brain through the use of neural-injury blood biomarkers, functional, diffusion, and perfusion MRI, and ocular-motor function across 3 time points (baseline, post-choking, post-non-choking). The central hypothesis is that acute neuronal structural, physiological, and functional alterations will be amplified after an incidence of choking-involved sex. The neural-injury blood biomarkers neurofilament light (NfL), glial fibrillary acidic protein (GFAP), Ubiquitin C-Terminal Hydrolase L1 (UCH-L1), and Tau will be measured in plasma, with the hypothesis that having choking involved sex will result in a increased heightened response compared to baseline and post non-choking involved sex timepoints. An additional panel of inflammatory cytokines may be considered if/when brain injury biomarkers show changes. It is also hypothesized that engaging in choking-involved sex will be associated with changes in fMRI activation patterns. White matter microstructure will be measured by diffusion imaging metrics, with the hypothesis that engaging in choking-involved sex will significantly disrupt microstructure at a post-choking involved sex time point, compared to baseline, but not at the post non-choking involved sex timepoint. The study will also assess oculomotor function as measured by near-point-of-convergence (NPC) in response to engaging in choking involved sex. The hypothesis is that NPC performance will be significantly impaired at the post choking-involved sex timepoint in comparison to both baseline and non-choking involved sex timepoints.

DETAILED DESCRIPTION:
The researchers will use a randomized controlled trial design and recruit participants on a first-come, first-serve basis for the study. This will be a crossover study where subjects will experience the same research interactions and data collection methods. Path 1 will involve 3 data collection time points including baseline data collection, post choking involved sex data collection time point, and post non-choking involved sex time point, in that order. Path 2 will involve 3 data collection time points including baseline data collection, post non-choking involved sex time point, and post choking involved sex time point, in that order. Each data collection timepoint will take approximately 2 hours. After enrollment, subjects will be sent a brief Qualtrics survey link once a day to determine when they are eligible for data collection based on their sexual activity within the last 24 hours. If a subject is eligible for data collection, they will come in on the following day.

When written informed consent is obtained, the researchers will use a self-reported health questionnaire to obtain demographic information. The information includes age, sex, romantic relationship status, sexual behavior habits, number and age of previous concussions, as well as assessment of other neurological conditions, psychosis screening, and MRI contradictions to screen participants' eligibility. Participants who meet the inclusion criteria and are free of exclusionary factors will advance to the testing procedures.

Enrollment Questionnaire:

The researchers will asses (1) impulsive behavior using SUPPS-P; (2) Childhood trauma load using CTQ; (3) lifetime trauma load using LEC5; (4) ADHD symptoms using WHO ASRS for DSM-5; (5) aggression in relationships using CTS2S; (6) insomnia symptoms using ISI, (7) migraine disability in the last 3 months using MIDAS (8) sex & sex behavior habits; (9) lifetime choking history; (10) lifetime sexual smothering/slapping history; (11) demographics; (12) alcohol use disorder using AUDIT; (13) cannabis use disorder using CUDIT; (14) MRI contradictions using MRI safety screening form

Data Collection Questionnaires:

The researchers will assess (1) depression, anxiety, perceived stress symptoms using the PHQ-9, GAD-7, and the Perceived Stress Scale; (2) neurobehavioral symptoms using the Neurobehavioral Symptom Inventory; (3) menstrual cycle; (4) health and behaviors in the last 24 hours related to sleep, head impacts, caffeine intake exercise, medication; (5) recent masturbation; (6) event level choking/slapping history

NPC:

During each test session, NPC assessment will be conducted on each participant. Near point of convergence (NPC) will be used to assessed ocular-motor function. The NPC measures the closest point to which one can maintain convergence while focusing on an object before double vision occurs. Assessment will be repeated twice, and mean NPC scores will be used for statistical analyses.

Blood Biomarkers:

Antecubital vein blood draws will be performed each test session to help determine serum biomarker concentrations. A trained phlebotomist will thoroughly clean the inner elbow surface with an alcohol swab and draw 7 ml of whole blood into sterile Vacutainer tubes with 21G butterfly needle. After the blood draw, the participant will use gauze to maintain direct pressure and a bandage will be provided. Plasma will be assessed by the 4-plex Simoa assay platform (Quanterix), which is a magnetic bead-based ELISA that allows detection of biomarkers in femtomolar concentrations. Additional panels of inflammatory cytokines/chemokines will be assessed by the Luminex system.

MRI Techniques:

Once completing the MRI screening procedure, participants will undergo the following standardized MRI protocols.

Diffusion tensor imaging (DTI): DTI is the most widely used technique to study the microstructural integrity of white matter in vivo. DTI provides simple markers, such as mean diffusivity (MD) and fractional anisotropy (FA), that have been used to reflect microstructural tissue change during aging, neurological disorders, and traumatic brain injury (i.e., concussion). However, despite their sensitivity, MD and FA represent cellular diffusivity estimated by basic statistical descriptions that do not directly correspond to biophysiological parameters of the neural cellular integrity. DTI assumes Gaussian diffusion within a single microstructural compartment and thus has proven non-specific to axonal structural damage. To address this limitation, neurite orientation dispersion and density imaging (NODDI) has been characterized to assess microstructural integrity of axons using a non-Gaussian model with multiple compartments. NODDI allows researchers to measure axonal density within white matter, orientation of axonal dispersion, and free water diffusion. The combined approach using NODDI and DTI will uncover greater depth of progressive axonal degeneration in response to sexual choking.

Perfusion: ASL (arterial spin labeling) MRI is an emerging non-invasive technique used to measure cerebral blood flow. ASL creates an image of blood flow throughout the brain by magnetically labeling blood water molecules as an intrinsic tracer while they travel to the brain. ASL offers an advantage over contrast bolus techniques as it is non-invasive and does not require the use of a contrast agent. Additionally ASL allows for the quantification of cerebral blood flow which offers an advantage over traditional contrast MR perfusion. The use of ASL MRI will uncover potential alteration in cerebral blood flow in response to sexual choking.

Resting-state fMRI: Measures of functional connectivity will be computed using a seed-based, correlational approach adapted for cortical surface-based analysis. The dorsolateral prefrontal cortex is set as our primary seed region, but all other regions (e.g., corpus callosum, angular gyrus, cingulate gyrus) will also be tested. Pre-analysis processing, surface sampling, ROI averaging, and motion censoring are adapted from the ABCD protocol. For network analysis, the investigators will calculate correlation values for each pair of ROIs, which are Fisher-transformed to z-statistics and averaged within or between networks to provide summary measures of network strength. The investigators will compute network metrics using the brain connectivity toolbox and compare connectivity measures within and between groups at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the age of 18-30
* Proficient in English
* Reports engaging in sex involving being choked at least 2 times in the past month

Exclusion Criteria:

* Pregnant
* History of moderate to severe TBI
* Has had a concussion in the last 6 months
* Any MRI contraindication (metal inside body near neck, face, head; metal IUD; severe claustrophobia; etc)
* Neurological condition (epilepsy, neurodegenerative disease, aneurysm, tumor, SCI, etc)
* Reports experiencing psychotic symptoms as measured by the Revised Behavior and Symptom Identification Scale
* Reports currently taking antipsychotic medication
* Reports less than 2 instances of being choked during partnered sexual events during the past month
* Reports engaging in sex without choking no times in the past month (i.e. reports strictly engaging in sex involving choking in the past month)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in brain-derived blood biomarkers from baseline to post choking involved sex time point | Blood samples will be collected at baseline and within 24 hours after engaging in sex involving choking
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), tau, and Ubiquitin C- terminal Hydrolase 1 (UCH-L1). All expression levels in pg/mL.
Differences in brain-derived blood biomarkers between post choking involved sex time point and post non-choking involved sex time point | Blood samples will be collected within 24 hours after engaging in sex involving choking and within 24 hours of engaging in non-choking involved sex
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), tau, and Ubiquitin C- terminal Hydrolase 1 (UCH-L1). All expression levels in pg/mL.
Differences in regional fMRI activation between post choking involved sex time point and post non-choking involved sex time point | fMRI procedures will be performed within 24 hours after engaging in sex involving choking and within 24 hours of engaging in non-choking involved sex
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to collect fMRI images while a risk taking task is administered.
  The task based fMRI protocol will consist of BART task to assess risk taking behavior and a function Resting State task.
Change in axonal microstructure from baseline to post choking involved sex time point | MRI procedures will be performed at baseline and within 24 hours after engaging in sex involving choking
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
Differences in axonal microstructure between post choking involved sex time point and post non-choking involved sex time point | MRI procedures will be performed within 24 hours after engaging in sex involving choking and within 24 hours of engaging in non-choking involved sex
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
Change in cerebral blood flow from baseline to post choking involved sex time point | MRI procedures will be performed at baseline and within 24 hours after engaging in sex involving choking
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in perfusion metrics.
Difference in cerebral blood flow between post choking involved sex time point and post non-choking involved sex time point | MRI procedures will be performed within 24 hours after engaging in sex involving choking and within 24 hours of engaging in non-choking involved sex
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in perfusion metrics.
Change in regional fMRI activation at rest from baseline to post choking involved sex time point | fMRI procedures will be performed at baseline and within 24 hours after engaging in sex involving choking
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to collect fMRI images while at rest.

SECONDARY OUTCOMES:
Change in ocular-motor function from baseline to post choking involved sex time point | Near point of convergence will be assessed at baseline and within 24 hours after engaging in sex involving choking
  Participants will undergo a brief test of near-point of convergence
Difference in ocular-motor function between post choking involved sex time point and post non-choking involved sex time point | Near point of convergence will be assessed within 24 hours after engaging in sex involving choking and within 24 hours of engaging in non-choking involved sex
  Participants will undergo a brief test of near-point of convergence

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be included in publications.

REFERENCES:
- [Background] Hou J, Huibregtse ME, Alexander IL, Klemsz LM, Fu TC, Rosenberg M, Fortenberry JD, Herbenick D, Kawata K. Structural brain morphology in young adult women who have been choked/strangled during sex: A whole-brain surface morphometry study. Brain Behav. 2023 Aug;13(8):e3160. doi: 10.1002/brb3.3160. Epub 2023 Jul 17. PMID 37459254
- [Background] Herbenick D, Fu TC, Eastman-Mueller H, Thomas S, Svetina Valdivia D, Rosenberg M, Guerra-Reyes L, Wright PJ, Kawata K, Feiner JR. Frequency, Method, Intensity, and Health Sequelae of Sexual Choking Among U.S. Undergraduate and Graduate Students. Arch Sex Behav. 2022 Aug;51(6):3121-3139. doi: 10.1007/s10508-022-02347-y. Epub 2022 Jul 28. PMID 35902430
- [Background] Hou J, Huibregtse ME, Alexander IL, Klemsz LM, Fu TC, Fortenberry JD, Herbenick D, Kawata K. Association of Frequent Sexual Choking/Strangulation With Neurophysiological Responses: A Pilot Resting-State fMRI Study. J Neurotrauma. 2023 Jul;40(13-14):1339-1351. doi: 10.1089/neu.2022.0146. Epub 2023 Feb 28. PMID 36565025
- [Background] Herbenick D, Fu TC, Patterson C, Rosenstock Gonzalez YR, Luetke M, Svetina Valdivia D, Eastman-Mueller H, Guerra-Reyes L, Rosenberg M. Prevalence and characteristics of choking/strangulation during sex: Findings from a probability survey of undergraduate students. J Am Coll Health. 2023 May-Jun;71(4):1059-1073. doi: 10.1080/07448481.2021.1920599. Epub 2021 Jul 9. PMID 34242530